CLINICAL TRIAL: NCT02124512
Title: Dietary Fat, Lipoprotein and Lipopolysaccharide: Role in Insulin Resistance
Brief Title: Blood Lipopolysaccharide (LPS) Rifaximin Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Sponsor-Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0136-F1V; UL1TR000117 (NIH); 1R21DK100258-01A1 (NIH)
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Obese; Insulin Resistance; Metabolic Syndrome
Keywords: obese; insulin resistance; metabolic syndrome
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Rifaximin SSD (Experimental): Subjects randomized to this arm of the study will receive 80 mg per day Rifaximin SSD
  Interventions: Drug: Rifaximin SSD
- Arm 2 Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifaximin SSD — Study Drug dosing will be 80 mg SSD once daily
  Arms: Arm 1 Rifaximin SSD
Other: Placebo — 80 mg placebo once daily
  Arms: Arm 2 Placebo

SUMMARY:
Metabolic syndrome is a condition involving elevated levels of fat in the blood, a tendency towards diabetes, hypertension, and too much fat around the abdomen (an increased waistline). Individuals with metabolic syndrome often have impaired glucose tolerance, which is a condition where blood sugar is normal when fasting (before eating), but is too high after drinking a sugary drink. This is due to an abnormality in the body's sensitivity to insulin (insulin resistance), which is due in part to an inability of the muscle to take up glucose.

People with metabolic syndrome have inflammation in their fat tissue and in their blood stream, and the changes in the level of inflammatory chemicals produced by cells in your fat tissues will be studied. One possible source of the inflammation may be the bacteria in the intestine. When individuals eat fatty foods, some of the bacterial products become attached to the fat in their blood and then get directed to fat tissue. The investigators wish to determine whether individuals have an excessive amount of inflammation in their fat tissues, and whether this inflammation comes from the bacteria in their intestines. To determine this, the investigators wish to treat individuals with an antibiotic that reduces the bacteria in their intestines and in their blood, and determine whether this reduces their overall level of inflammation.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled proof of concept study that will examine the investigational drug Rifaximin Soluble Solid Dispersion (SSD) ability to reduce gut microbiota and thereby reduce adipose inflammation and improve insulin resistance.

Each subject enrolled will undergo a fat tolerance test with a high-fat meal, an oral glucose tolerance test, a fat biopsy, and a euglycemic clamp. Following their successful completion of those procedures subjects will be randomized to study treatment. That treatment will involve receiving the investigational drug,80 mg per day of rifaximin-soluble solid dispersion (SDD), or placebo for 12 weeks. All procedures will be performed on the Clinical Services Core of the CCTS. The initial visit will involve informed consent, and routine labs (comprehensive metabolic panel, lipid panel, TSH, CBC with platelets). These routine labs are for safety purposes and to rule out exclusionary disorders. A stool sample will also be collected and frozen for possible future analysis of bacterial microflora.

Subjects will be asked to allow the principal investigator to bank blood and tissue samples collected during this study that are not used for other study-related tests. No additional blood or tissue samples will be collected. If the subject agrees to the banking of their blood and tissue samples they will be stored in the Principal Investigator's laboratory at the University of Kentucky for an indefinite period of time or until they are used up. Stored samples will be used for future research testing to learn about how to prevent, detect, or treat insulin resistance, metabolic syndrome, diabetes or other health problems.

Each subject will undergo total body composition testing using a total body dual-energy x-ray absorptiometry (DXA) scan. The DXA scan measures the subject's bond density and body fat.

ELIGIBILITY:
Inclusion Criteria:

* Obese
* Insulin resistance or metabolic syndrome
* Body Mass Index between 27 and 45
* Waist circumference >40" (M) or >35" (F)
* Impaired glucose tolerance (IGT)
* Normal glucose tolerance (NGT) with at least three features of MetS
* A1C <6.5
* Blood pressure 130/85

Exclusion Criteria:

* Pregnant or breastfeeding
* Recent or unstable cardiovascular disease
* cancer,
* Renal insufficiency (GFR<30)
* Steroid use
* chronic inflammatory conditions
* Anticoagulant use
* Lipodystrophy
* Irritable Bowel Syndrome
* Allergy to local anesthetic
* Lactose intolerance

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phililp Kern, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Center for Clinical and Translational Science, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 Rifaximin SSD | Arm 2 Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Rifaximin SSD | Arm 2 Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (3.0) | 50 (2.9) | 50 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 38.5 (4.2) | 36.1 (3.4) | 37.3 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Circulating LPS
Description: Plasma lipopolysaccharide (LPS) will be measured both in the fasting state and after a lipid-rich meal in obese subjects (Pre-Treatment: 0, 4 and 8 hr timepoints). The subjects will then be treated with the antibiotic rifaximin for 12 weeks to substantially reduce gut bacteria. LPS measurements at fasting and after a lipid-rich meal will be repeated (Post-Treatment: 0, 4 and 8 hr timepoints). The lipid tolerance tests before and after treatment with rifaximin will be assessed to determine whether there is a reduction in post-prandial LPS. LPS measurements were obtained using a modified LAL Assay.
Time Frame: 0, 4 and 8 hours at Baseline, and 0, 4 and 8 hours after 12 weeks of treatment
Measure: Mean (Standard Error); unit: EU/mL
Arm/Group | Arm 1 Rifaximin SSD | Arm 2 Placebo
Number analyzed (Participants) | 6 | 6
EU/mL
  Pre-treatment 0hr | 2.44 (0.40) | 1.86 (0.33)
  Pre-treatment 4hr | 13.66 (2.93) | 10.00 (1.55)
  Pre-treatment 8hr | 1.71 (0.26) | 1.04 (0.48)
  Post-treatment 0hr | 1.89 (0.35) | 1.86 (0.43)
  Post-treatment 4hr | 8.45 (1.87) | 9.97 (4.30)
  Post-treatment 8hr | 2.14 (0.49) | 2.29 (0.81)
Statistical Analysis 1: Comparison: Arm 1 Rifaximin SSD vs Arm 2 Placebo; Comparison of the pre- and post-treatment timecourse between untreated and rifaximin-treated participants; Test type: Superiority; p > 0.05, ANOVA — The p-value was calculated to be >0.05

2. Secondary Outcome: Tissue Inflammation
Description: Subjects will undergo a baseline fat biopsy (pre-treatment). They will then be treated with rifaximin for 12 weeks and biopsies will be repeated to determine if disruption of the microbiota reduces tissue inflammation. Data are reported as normalized mRNA expression levels (arbitrary units) of TNFalpha.
Time Frame: Pre-Treatment (baseline) and Post-Treatment (12 weeks after baseline).
Measure: Mean (Standard Error); unit: arbitrary units
Arm/Group | Arm 1 Rifaximin SSD | Arm 2 Placebo
Number analyzed (Participants) | 6 | 6
arbitrary units
  Pre-Treatment | 2.00 (0.25) | 1.30 (0.13)
  Post-Treatment | 1.67 (0.25) | 1.46 (0.28)
Statistical Analysis 1: Comparison: Arm 1 Rifaximin SSD vs Arm 2 Placebo; Treatment difference (change in placebo pre- and post-treatment versus change in rifaximin pre- and post-treatment); Test type: Superiority; p = 0.12, t-test, 2 sided — unpaired Student's t-test

3. Other Pre Specified Outcome: Improved Insulin Sensitivity
Description: We hypothesize that a change in the microbial flora with rifaximin will alter plasma LPS, adipose tissue inflammation, and insulin sensitivity. Therefore, we will examine, before and after rifaximin/placebo treatment: 1. LPS associated with lipoproteins, 2. insulin sensitivity and hepatic glucose production, 3. plasma inflammatory markers (TNFα, IL-6, MCP-1, adiponectin), 4. adipose inflammatory markers (CD68, MCP1, TNFα, PAI1, IL12, IL10, TLR4 and others).
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Arm 1 Rifaximin SSD | Arm 2 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02124512/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02124512/ICF_001.pdf